CLINICAL TRIAL: NCT03904992
Title: Intervention With a Progressive Web App for the Promotion of Healthy Habits in Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 102342
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Health Behavior
Keywords: Nutrtition; Physical activity; Preescholer; Informatics
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: First, a baseline evaluation will be made to the participants, based on the indicators of interest.
  During a period of 60 days, the caregivers of the intervention group had free access to the progressive web app "Nutrinidos" and received training for its use. On the other hand, nutritional counseling was available every 30 days for the participants assigned to the control group. They consisted of personalized sessions with a duration of 20 minutes in which parents and caregivers could resolve their doubts regarding the feeding of their children. In addition, they were offered physical education materials designed and adapted with content used in this study. The educational material addressed contains information about lunch boxes, eating habits, consumption of fruits and vegetables, prevention of anemia, and physical activity.
  After 60 days of follow-up, the evaluation of results will be carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-exposed (No Intervention): Subjects with access to nutritional counseling sessions every 30 days
- Exposed (Experimental): Subjects with access to the progressive web app in their smartphones.
  Interventions: Other: Progressive web app

INTERVENTIONS:
Other: Progressive web app — Access to a progressive web app for the promotion of healthy habits in preescholers through the participant's smatphone
  Arms: Exposed

SUMMARY:
The preschool stage has been identified as an important moment for the study of factors associated with obesity. The worrying national situation of overweight in children from 3 to 5 years old, the increase in consumption of ultra-processed foods nationwide that is associated with the increase of the body mass index at the national level, the reduced national scientific evidence regarding the effectiveness of interventions in promoting healthy habits, as well as the lack of tools for mothers of preschool children in nutrition and physical activity, make interventions necessary in this area. On the other hand, currently, users worldwide are installing fewer applications and, although they spend more time using mobile applications, they are limited to a handful. Therefore, developing a native mobile application that is highly consumed is very difficult and expensive. For this reason, progressive web apps emerge as an attractive alternative for users given its attractive features, cross-platform interface, lower development cost and a growing demand for such applications. Thus, this research seeks to explore a novel way to promote healthy habits in preschoolers and check their effectiveness. In this way, a precedent could be set in the use of technologies in health promotion that could be extended to other age groups.

DETAILED DESCRIPTION:
SAMPLE SIZE The sample size was calculated using OpenEpi (www.openepi.com), with the sample size formula to compare two means, considering a confidence interval of 95%, power of 80%, ratio of sample size (group 2 / group 1) equal to 1, a minimum expected mean difference of 5 points and a standard deviation of 9.5 points for both groups. Thus, the required sample size is 114 participants (57 intervened and 57 not intervened).

TECHNIQUES AND PROCEDURES FOR DATA COLLECTION

First stage: Design of the progressive web app

In this phase, the profile of the users will be defined through a focus group. Among the information gathered is socio-demographic data, use of technology, current situation of the feeding and physical activity of the preschool, and expectations of the functions of the computer tool. In addition, a complementary bibliographic search will be carried out on the subject to expand the information necessary for the design of the PWA.

Based on the information collected, the alpha version of the application will be developed. It will undergo a validation process and based on the feedback, the application will be improved until a beta version is developed.

Second stage: intervention with the progressive web app (PWA)

ANALYSIS PLAN

The data was collected using the Magpi software. To verify the comparability of the two randomization groups based on the sociodemographic covariates through a descriptive analysis, a frequency and percentage table was constructed, which were compared by statistical tests.

In addition, the variation of the ration consumption of the food groups, the score in each component of the feeding behavior and the activity of the preschool was analyzed; the variation of the nutritional status and quality of the components of the lunch box in the control and intervention group was identified; and the variation of the Z score for the indicator of BMI for age and the consumption of the lunch box was plotted through a chart of boxes.

To determine the effect of the intervention, the differences of the measurements (post-pre) of the control and intervention groups were compared. For this, the Student t test was used for independent samples. The variables analyzed were:

* Variation of the dietetic quality of the preschool
* Variation in the nutritional status of children
* Variation of preschool feeding behavior
* Variation of the composition of the lunchbox
* Variation of the consumption of the lunchbox
* Variation of physical activity Finally, a satisfaction survey was applied to the intervention group and the results were presented using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children from 3 to 6 years old that currently attend school
* People who have access to a mid-range or high-end Smartphone with Android 6.0 operating system or higher, with Internet access, in which the application will be installed

Exclusion Criteria:

* Caregivers of children with hormonal diseases that affect the nutritional status (referred by caregiver or caregiver): hypothyroidism, hyperthyroidism, Cushing's syndrome, growth hormone deficiency, diabetes
* Caregivers of children with heart disease, kidney disease or cancer (referred by caregiver or caregiver)
* Caregivers of children with paraplegia, tetraplegia or some degree of paralysis
* Caregivers of children who are beneficiaries of the Qali Warma Program
* People who are illiterate or who have great difficulties in the operation of smartphones

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Variation of the dietary diversity of the preescholer | 60 days after the instalation of the Progressive Web App
  The difference between the scores obtained in the baseline and the evaluation using the Healthy Eating Index score

SECONDARY OUTCOMES:
Variation in preescholer's nutritional status | 60 days after the instalation of the Progressive Web App
  The difference between the Z-point values of the BMI for age pattern.
Variation of the preescholer's eating behavior | 60 days after the instalation of the Progressive Web App
  The difference between the scores obtained for child's eating behavior that will be evaluated through the Children Eating Behaviour Questionnaire
Variation of the composition of the lunch box | 60 days after the instalation of the Progressive Web App
  Change in the score obtained for the composition of the preescholer's lunch boxes
Variation of the refreshment consumption | 60 days after the instalation of the Progressive Web App
  The change in the consumption of the refreshments (lunch box) will be determined using a food scale (grams).
Variation of physical activity | 60 days after the instalation of the Progressive Web App
  A difference in the number of minutes of physical activity of the preschoolers reported by the parents using a validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Oscar J Calvo Torres, BS, Principal Investigator
Locations (1):
- I.E.I. Juan Pablo Peregrino, San Martín de Porres, Lima region, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Revilla L, Alvarado C, Álvarez D, Tarqui C, Gómez G, Jacoby E, et al. Un gordo problema: Sobrepeso y Obesidad en el Perú. Editor Imprenta Sanchez SRL [Internet]. 2012;1-24. Available from: http://bvs.minsa.gob.pe/local/MINSA/1830.pdf
- [Background] Tarqui C, Sánchez J, Alvarez D, Gómez G, Valdivia S. Tendencia del sobrepeso, obesidad y exceso de peso en el Perú. La Rev Peru Epidemiol [Internet]. 2013;17(3):7. Available from: http://ateneo.unmsm.edu.pe/ateneo/bitstream/123456789/3132/3/rev_peru_epidemiol04v17n3_2013.pdf%5Cnhttp://rpe.epiredperu.net/rpe_ediciones/2013_v17_n03/Original tendencia del sobrepeso y obesidad en Peru RPE 17_3.pdf
- [Background] Instituto Nacional de Salud. Situación Nutricional - Obsevatorio de Nutrición y el Estudio del Sobrepeso y Obesidad [Internet]. [cited 2018 Apr 18]. Available from: http://www.observateperu.ins.gob.pe/sala-situacional/situacion-nutricional
- [Background] Ruiz EF, Proano A, Ponce OJ, Curioso WH. [Mobile health for public health in Peru: lessons learned]. Rev Peru Med Exp Salud Publica. 2015 Apr-Jun;32(2):364-72. Spanish. PMID 26338384
- [Background] Santiago MA, Fernández RN, Esquirol JRL, Sánchez IP. La edad preescolar como momento singular del desarrollo humano. Rev Cubana Pediatr. 2007;79(4) Available from: http://www.aeped.es/documentos/protocolos-nutricion
- [Background] Rojas A, León M, Sánchez O. Formación de hábitos alimentarios y de estilos de vida saludables. Curric Educ Inicial [Internet]. 2003;1-36. Available from: http://www.unicef.org/venezuela/spanish/educinic9.pdf
- [Background] Pediatría C de N de la SU de. Guías de alimentación del niño preescolar y escolar. Arch Pediatr Urug. 2004;75(2):159-13.
- [Background] Cortina LS. Protocolos de nutrición. Protoc la AEP [Internet]. 2010;297-305. Available from: http://www.aeped.es/documentos/protocolos-nutricion
- [Background] Trost SG, Sirard JR, Dowda M, Pfeiffer KA, Pate RR. Physical activity in overweight and nonoverweight preschool children. Int J Obes Relat Metab Disord. 2003 Jul;27(7):834-9. doi: 10.1038/sj.ijo.0802311. PMID 12821970
- [Background] Gmbh GG, Steiner T. What is in a Web View ? An Analysis of Progressive Web App Features When the Means of Web Access is not a Web Browser. In: Companion of the The Web Conference 2018 on The Web Conference 2018. Ginebra, Suiza: International World Wide Web Conferences Steering Committee; 2018. p. 789-96.
- [Background] Ater T. Building Progressive Web Apps: Bringing the Power of Native to the Browser. 1ed ed. EE.UU.: O'Reilly Media; 2017. 288 p.
- [Background] Sheppard D (Computer software developer). Beginning progressive web app development creating a native app experience on the web [Internet]. EE.UU.: Apress Media LLC; 2017. Available from: https://books.google.mu/books?id=9_RADwAAQBAJ&dq=progressive+web+apps&source=gbs_navlinks_s
- [Background] OPS. Alimentos y bebidas ultraprocesados en América Latina: tendencias, efecto sobre la obesidad e implicaciones para las políticas públicas [Internet]. Washington D.C.: Organización Panamericana de la Salud; 2015 [cited 2018 Apr 30]. Available from: http://iris.paho.org/xmlui/bitstream/handle/123456789/7698/9789275318645_esp.pdf
- [Background] Leal KK, Schneider BC, Franca GV, Gigante DP, dos Santos I, Assuncao MC. [Diet quality of preschool children aged 2 to 5 years living in the urban area of Pelotas, Brazil]. Rev Paul Pediatr. 2015 Jul-Sep;33(3):311-8. doi: 10.1016/j.rpped.2015.05.002. Epub 2015 Jun 10. PMID 26122208
- [Background] Rauber F, da Costa Louzada ML, Vitolo MR. Healthy eating index measures diet quality of Brazilian children of low socioeconomic status. J Am Coll Nutr. 2014;33(1):26-31. doi: 10.1080/07315724.2014.869979. PMID 24533605
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Zelenko O, Tjondronegoro D, Mani M. Mobile app rating scale: a new tool for assessing the quality of health mobile apps. JMIR Mhealth Uhealth. 2015 Mar 11;3(1):e27. doi: 10.2196/mhealth.3422. PMID 25760773
- [Background] Carbajal I. Estado nutricional y consumo de energía y nutrientes en un grupo de adolescentes de Lima y Callao. Universidad Nacional Mayor de San Marcos; 2001.
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Carnell S, Wardle J. Measuring behavioural susceptibility to obesity: validation of the child eating behaviour questionnaire. Appetite. 2007 Jan;48(1):104-13. doi: 10.1016/j.appet.2006.07.075. Epub 2006 Sep 7. PMID 16962207
- [Background] Camargo DM, Santisteban S, Paredes E, Florez MA, Bueno D. [Reliability of a questionnaire for measuring physical activity and sedentary behavior in children from preschool to fourth grade]. Biomedica. 2015 Jul-Sep;35(3):347-56. doi: 10.7705/biomedica.v35i3.2502. Spanish. PMID 26849696
- [Background] Organización Mundial de la Salud. Interpretando los Indicadores de Crecimiento Interpretando los Indicadores [Internet]. Curso de Capacitación sobre la Evaluación del Crecimiento del Niño. 2008. 56 p. Available from: http://www.who.int/childgrowth/training/c_interpretando.pdf